CLINICAL TRIAL: NCT02536196
Title: A Randomized Evaluation of the TriGuard Embolic Deflection Device to Reduce the Impact of Cerebral Embolic Lesions After Transcatheter Aortic Valve Implantation
Brief Title: The REFLECT Trial: Cerebral Protection to Reduce Cerebral Embolic Lesions After Transcatheter Aortic Valve Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keystone Heart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REFLECT
Record Dates: First submitted 2015-08-26; First posted 2015-08-31 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Symptomatic Aortic Stenosis
Keywords: Aortic stenosis; TAVI; TriGUARD; Keystone Heart; Cerebral Embolic Protection
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Embolic Protection Devices; Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Embolic Protection with transcatheter aortic valve implantation (TAVI)
  Interventions: Device: Embolic Protection Device; Procedure: Transcatheter aortic valve implantation (TAVI)
- Control Arm (Active Comparator): Transcatheter aortic valve implantation (TAVI) without embolic protection
  Interventions: Procedure: Transcatheter aortic valve implantation (TAVI)

INTERVENTIONS:
Device: Embolic Protection Device — Embolic protection
  Arms: Intervention
Procedure: Transcatheter aortic valve implantation (TAVI) — Transcatheter aortic valve implantation (TAVI)

SUMMARY:
The Keystone Heart TriGuard™ HDH is an aortic embolism deflection device intended to reduce the amount of embolic material that may enter the carotid, subclavian, and vertebral arteries during transcatheter heart valve implantation.

The objective of the study is to assess the safety and efficacy of the TriGuard™ HDH embolic deflection device in patients undergoing transcatheter aortic valve implantation (TAVI), in comparison with an active control group of patients undergoing unprotected TAVI.

Subjects with indications for TAVI and who meet study eligibility criteria will be randomized 2:1 to one of two treatment arms: 1) Intervention: Embolic protection device (TriGuard™) with transcatheter aortic valve implantation or 2) Control: Unprotected transcatheter aortic valve implantation.

DETAILED DESCRIPTION:
This prospective, single-blind, three arm, randomized, (2 device: 1 control), multicenter safety and efficacy trial is designed to enroll up to 603 total subjects in two consecutive phases: Phase I enrolled 258 subjects (including 54 Roll-Ins) and utilized the TriGuard HDH and Phase II will enroll up to 345 subjects (including 40-50 Roll-Ins) and will utilize the TriGUARD 3 (Figure 3b shows the patient flow/disposition).

Phase I In phase I, a total of 204 evaluable subjects and 54 roll-in subjects were enrolled at 26 total investigational sites in the United States, Europe, and Israel, of which 20 sites were in the United States. A minimum of 50% of subjects were planned to be enrolled at US sites, and no single site was permitted to enroll more than 20% of all subjects.

Subjects with indications for TAVI and who met study eligibility criteria were randomized 2:1 (stratified by study site) to one of two treatment arms:

* Intervention (Phase 1 Cohort) - TAVI with the TriGuard HDH CEPD
* Control - standard unprotected TAVI At sites where the investigator did not have prior experience with the TriGuard device (minimum of 2 prior cases), up to 3 roll-in subjects were enrolled. Roll-in subjects were not randomized, but underwent TAVI with the TriGuard HDH device. These cases were proctored by a Sponsor representative. Investigational sites with ≥2 prior TriGuard cases were allowed to enroll 1 roll-in subject at the discretion of the site principal investigator.

All subjects were to be followed clinically in-hospital and at 30 and 90 days, and to undergo diffusion-weighted MR imaging 2 to 5 days post-procedure, and neurologic and neuropsychological testing pre-procedure, post-procedure (2-5 days post-procedure), and at 30 and 90 days.

The initial randomized cohort expected to enroll up to 285 subjects. Note: Enrollment in Phase I has been halted after enrolling a total of 258 subjects (54 roll-ins and 204 randomized subjects including 63 controls) based on the recommendation of the Data Monitoring Committee following a review of interim 30-day data on 90 subjects at the prespecified interim analysis time point. A next iteration device designed for increased efficacy, ease of use, and improved safety will be tested in Phase II (below).

Phase II In Phase II, up to 295 randomized subjects and 40-50 roll-in subjects will be enrolled at up to 25 sites in the United States (inclusive of sites enrolling subjects in Phase I). No single site will be permitted to enroll more than 20% of all randomized subjects in Phase II.

Subjects with indications for TAVI and who meet study eligibility criteria will be randomized 2:1 (stratified by study site) to one of two treatment arms:

* Intervention - TAVI with the TriGUARD 3 CEPD
* Control - standard unprotected TAVI. Randomization will be stratified by implanted valve type (Medtronic vs. Edwards).

No single valve type will be implanted in more than approximately 70% of randomized patients (phase II).

Roll-in subjects (a minimum of 2 and a maximum of 3 Roll-ins per-site) will not be randomized, but will undergo TAVI with the TriGUARD 3 device. These cases will be proctored by a Sponsor representative.

All subjects will be followed clinically in-hospital and at 30 days, undergo diffusion-weighted MR imaging 2 to 5 days post-procedure, and undergo neurologic (NIHSS) testing pre-procedure, post-procedure (2-5 days post-procedure), and at 30 days. A follow-up phone-call to assess the occurrence of death or stroke will be done at 90 days.

The initial randomized cohort will consist of up to 225 subjects. After at least 50% of the initial randomized cohort (approximately 112 subjects) have reached the 30 day primary efficacy endpoint evaluation time point, a sample size reestimation will be performed in case the conditional power of the trial (assessed by the independent biostatistician) is >40% but <80%, subject to approval by the Sponsor. If this analysis determines that more than 225 randomized subjects will be required to ensure adequate study power, enrollment may continue until the required number of subjects have been enrolled, or until the total subject limit for the study has been reached (whichever occurs first).

ELIGIBILITY:
Subjects must meet ALL of the following criteria:

General Inclusion Criteria

1. The patient is a male or non-pregnant female ≥18 years of age
2. The patient meets indications for transcatheter aortic valve implantation (TAVI)
3. The patient is willing to comply with protocol-specified follow-up evaluations
4. The patient, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC).

Potential Subjects will be excluded if ANY of the following criteria apply:

General Exclusion Criteria

1. Patients undergoing transcatheter aortic valve implantation (TAVI) via the trans-axillary, trans-subclavian, or trans-aortic route
2. Patients undergoing transcatheter aortic valve implantation (TAVI) via the transapical approach due to friable or mobile atherosclerotic plaque in the aortic arch
3. Patients with a previously implanted prosthetic aortic valve (i.e., planned valve-in-valve transcatheter aortic valve implantation (TAVI))
4. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 14 days prior to index procedure per site standard test
5. Patients with known diagnosis of acute myocardial infarction (AMI) within 72 hours preceding the index procedure (according to definition) or AMI >72 hours preceding the index procedure, in whom Creatine Kinase (CK) and CK-MB have not returned to within normal limits at the time of procedure, or patients who are currently experiencing clinical symptoms consistent with new-onset AMI, such as nitrate-unresponsive prolonged chest pain
6. Patients with a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated, patients who will refuse transfusion, or patients with an active peptic ulcer or history of upper gastrointestinal (GI) bleeding within the prior 3 months
7. Patients with known mental or physical illness or known history of substance abuse that may cause non-compliance with the protocol, confound the data interpretation, or is associated with a life expectancy of less than one year
8. Patients with severe allergy or known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel, nitinol, stainless steel alloy, and/or contrast sensitivity that cannot be adequately pre-medicated
9. Patients with a history of a stroke or transient ischemic attack (TIA) within the prior 6 months
10. Patients with renal failure (estimated Glomerular Filtration Rate [eGFR] <30 mL/min, calculated from serum creatinine by the Cockcroft-Gault formula)
11. Patients with hepatic failure (Child-Pugh class C)
12. Patients with hypercoagulable states that cannot be corrected by additional periprocedural heparin
13. Patients presenting with cardiogenic shock at the time of the index procedure
14. Patients with severe peripheral arterial, abdominal aortic, or thoracic aortic disease that precludes delivery sheath vascular access
15. Patients in whom the aortic arch, innominate artery ostium, or proximal innominate artery is heavily calcified, severely atheromatous, or severely tortuous
16. Patients with an innominate artery ostium diameter <10 mm or >25 mm
17. Patients with a transverse aortic diameter >43
18. Patients with anatomic irregularities of the innominate artery that could prevent positioning of the TriGuard upper stabilizer and compromise stability of the device
19. Patients with any other condition that would prevent adherence to the TriGuard HDH Instructions for Use
20. Patients with contraindication to cerebral MRI
21. Patients who have a planned treatment with any other investigational device or procedure during the study period
22. Patients planned to undergo any other cardiac surgical or interventional procedure (e.g., concurrent coronary revascularization) during the TAVI procedure or within 10 days prior to the TAVI procedure. NOTE: Diagnostic cardiac catheterization is permitted within 10 day prior to the TAVI procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra J Lansky, MD, Principal Investigator — alexandra.lansky@yale.edu
Locations (30):
- United States (23):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Foundation for Cardiovascular Medicine, San Diego, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Delray Medical Center, Hialeah, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - University of Iowa, Iowa City, Iowa
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Morristown Medical Center, Morristown, New Jersey
  - New York University, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Pinnacle Health, Harrisburg, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor Heart and Vascular HospitalBaylor Heart and Vascular, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas, Houston, Texas
  - Baylor Research Center, Plano, Texas
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
- Germany (4):
  - University of Bonn, Bonn
  - Universitats-Herzzentrum Freiburg, Freiburg im Breisgau
  - Hamburg Univeristy Cardiovascular Center, Hamburg
  - Leipzig Heart Institute, Leipzig
- Italy (2):
  - San Donato Hospital, Milan
  - San Rafeele Hospital, Milan
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Lansky AJ, Grubman D, Dwyer MG 3rd, Zivadinov R, Parise H, Moses JW, Shah T, Pietras C, Tirziu D, Gambone L, Leon MB, Nazif TM, Messe SR. Clinical Significance of Diffusion-Weighted Brain MRI Lesions After TAVR: Results of a Patient-Level Pooled Analysis. J Am Coll Cardiol. 2024 Aug 20;84(8):712-722. doi: 10.1016/j.jacc.2024.05.055. PMID 39142725

RESULTS

PARTICIPANT FLOW:
Groups:
- Roll-in: These are patients that were the initial 2 to 3 patients per site that recieved the device but were used to train physicians but not in the randomized group
Period: Overall Study
Arm/Group | Intervention | Control Arm | Roll-in
Started | 262 | 121 | 95
Completed | 233 | 107 | 95
Not Completed | 29 | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- Roll-In: Embolic Protection with transcatheter aortic valve implantation (TAVI)
  Embolic Protection Device: Embolic protection
  Transcatheter aortic valve implantation (TAVI): Transcatheter aortic valve implantation (TAVI)
  Only used for training / safety. No efficacy measurements
- Total: Total of all reporting groups
Arm/Group | Intervention | Control Arm | Roll-In | Total
Number analyzed (Participants) | 262 | 121 | 95 | 478
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 2 | 7
  >=65 years | 259 | 119 | 93 | 471
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 44 | 44 | 199
  Male | 151 | 77 | 51 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 2 | 14
  Not Hispanic or Latino | 255 | 116 | 93 | 464
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 220 | 108 | 90 | 418
  Europe | 42 | 13 | 5 | 60
Prior CVA/TIA [Count of Participants; unit: Participants] | 38 | 10 | 14 | 62

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint - Composite Safety Endpoint Based on MACCE
Description: Combined safety endpoint at 30 days defined according to VARC-2 ("TAVI early safety") as a composite of:
  1. All-cause mortality - number of patients that expired
  2. All stroke (disabling and non-disabling) - defined by VARC-2 scale
  3. Life-threatening or disabled bleeding - BARC bleeding scale - 5 point scale ranging from no bleeding to fatal
  4. Acute kidney injury - Stage 2 or 3 (including renal replacement therapy)
  5. Coronary artery obstruction requiring intervention
  6. Major vascular complication, and
  7. Valve-related dysfunction requiring repeat procedure (BAV, TAVI, or SAVR) - number of patients in whom a valve related dysfunction occurred It was pre-specified to combine all participants that received the device in the andomized Intervention and Roll-in Arms/Groups for this Outcome Measure.
Time Frame: 30 Days
Population: The population that received the investigational device, Treatment and Rollin patients against safety performance goal. 5 patients withdrew prior to receiving the device resulting in 157 (121Tx+41RI-5). Control patients did not receive the device and were not evaluated in safety endpoint. Composite endpoint is comprised of the number of events against total number of events in accordance with MACCE. The safety endpoint was pre-specified to be calculated separately for the Roll-In population.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 157
Participants | 25

2. Primary Outcome: Primary Efficacy Endpoint
Description: Hierarchical composite efficacy endpt, determined by pair-wise comparisons among subjects according to hierarchy:
  * mortality or any stroke [30 days]
  * death/stroke time to event analysis by days determine win
  * stroke at same day the comparison moves to next tier
  * NIHSS worsening [2-5 days post]
  * Freedom from lesions detected by DW-MRI 2-5 days post
  * Total volume lesions detected by DW-MRI 2-5 days post Each subj in intervention compared with each subj from control based on hierarchy according to Finkelstein-Schoenfeld method. If Subj A dies or has stroke &Subj B survives free of stroke to 30 days, Subj B wins(score+1) &Subj A loses (score-1). Both die or have stroke, patient with later event wins. Both have death/stroke on same day is equilibrium (score 0). Both are alive & have stroke on same day, comparison moves to next tier. Both stroke-free to 30 days, comparison moves to the next tier. Scores summed to cumulative score for each subj, &outcomes between groups are compared.
Time Frame: Pre-discharge through 30-days
Population: eITT population consists of those patients that received the device, i.e. didn't withdraw prior to receiving the investigational device. Of 121 interventional patients in phase 2 of the protocol, 9 patients withdrew before receiving the device. From the total 121 control patients, 2 of the subjects withdrew before receiving the TAVI. There is no theoretical min and max as the number of events could not be known ahead of time, ROLL-IN PATIENTS ARE NOT INCLUDED IN THE EFFICACY ENDPOINT
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Without CEP
Arm/Group | Intervention | Control
Number analyzed (Participants) | 112 | 119
units on a scale | 587.8 (1028.42) | 508.2 (1123.96)

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Intervention: Embolic Protection with transcatheter aortic valve implantation (TAVI)
  Embolic Protection Device: Keystone Heart TriGUARD 3
- Control: The control group received a TAVI but did not receive a cerebral embolic protection device.
- Roll In: Patients who received the investigational device - TriGUARD 3 but were used for physician training.
Arm/Group | Intervention | Control | Roll In
All-Cause Mortality (participants affected / at risk) | 4/157 | 1/63 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/157 | 2/63 | 1/41
Other Adverse Events (participants affected / at risk) | 130/157 | 43/63 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=157) | Control (N=63) | Roll In (N=41)
Vascular Bleed (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) — vascular complications with closure; not directly related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=157) | Control (N=63) | Roll In (N=41)
Blood and Lymphatic (Blood and lymphatic system disorders) | 24 (29) | 7 (7) | 0
Cardiac (Cardiac disorders) | 83 (122) | 27 (35) | 0
General Disorders (General disorders) | 19 (19) | 4 (4) | 0
Infections and Infestations (Infections and infestations) | 13 (16) | 5 (5) | 0

LIMITATIONS AND CAVEATS:
Study sample size was limited and imbalance in cohorts / randomization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT02536196/Prot_SAP_000.pdf